CLINICAL TRIAL: NCT02705222
Title: Comparison Between Dilatation and Curettage and Hysteroscopy in Management of Abnormal Uterine Bleeding in Perimenopausal Women
Brief Title: Comparison Between D&C and Hysteroscopy in Management of AUB in Perimenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SMM
Record Dates: First submitted 2016-02-26; First posted 2016-03-10 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Uterine Bleeding
Keywords: Abnormal uterine bleeding; Dilatation and curettage; Hysteroscopy
MeSH Terms: conditions — Uterine Hemorrhage; Metrorrhagia; Dilatation, Pathologic | interventions — Dilatation and Curettage; Hysteroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D&C group (Active Comparator): Women will undergo D&C
  Interventions: Procedure: D&C
- Hysteroscopy group (Active Comparator): Women will undergo hysteroscopy
  Interventions: Procedure: Hysteroscopy

INTERVENTIONS:
Procedure: D&C — Cervical dilatation and fractional endometrial curettage will be done in operation theatre and the curetting will be sent for histopathological examination
  Other Names: Dilatation and curettage
  Arms: D&C group
Procedure: Hysteroscopy — Hysteroscopy will be done in operation theatre and hysteroscopic-guided curettings will also be taken and sent for histopathological examination
  Arms: Hysteroscopy group

SUMMARY:
The aim of this study is to compare dilatation and curettage with hysteroscopy in obtaining an accurate diagnosis of the etiology of abnormal uterine bleeding and outlining a mode of treatment-specific to the cause.

DETAILED DESCRIPTION:
Perimenopausal women complaining of abnormal uterine bleeding will be selected for assessment through detailed history taking, general and abdominal examination, local gynecological examination, transvaginal sonography (TVS) scanning and routine blood investigations. Eligible participants in our study will be those who complain of menorrhagia, metrorrhagia, polymenorrhoea or polymenorrhagia without local gynecological cause with failure of medical treatment for at least 3 months. All women participating in the study will be randomly allocated into two groups; dilatation and curettage (D&C) group and hysteroscopy group. For women in the D&C group, cervical dilatation and fractional endometrial curettage will be done under total intravenous (IV) anesthesia in operation theater and the curetting will be sent for histopathological examination. For women in the hysteroscopy group, hysteroscopy will be done under total IV anesthesia in operation theater hysteroscopic-guided curettings will also be taken and sent for histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women complaining of abnormal uterine bleeding (menorrhagia, metrorrhagia, polymenorrhoea or polymenorrhagia) without local gynecological cause.
* Failure of medical treatment for at least 3 months.

Exclusion Criteria:

* Age < 45 or > 55 years.
* Blood disorders or coagulopathy.
* Diagnosed or suspected local gynecologic lesion (polyp, adenomyosis, myoma, malignancy or cervical pathology).
* Use intrauterine contraceptive device.
* Pregnancy related conditions.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Percentage of abnormal endometrial patterns | One week after the procedure
  Number of patients diagnosed to have abnormal endometrial patterns after histopathological examination of the curretings per total number of patients underwent the procedure

SECONDARY OUTCOMES:
Improvement rate | 3 months after the procedure
  Number of patients improved after performing the procedure and recieving the treatment-specific to cause per total number of patients underwent the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Madany, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University; Moustafa H Nawwar, Dr, Study Director — Mansoura University; Mohamed A Elnegeri, Prof, Study Chair — Mansoura University
Locations (1):
- Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided